CLINICAL TRIAL: NCT00536887
Title: Phase 4 Study of Atorvastatin 10mg vs. 40mg in Follow-up CFR in AMI Patients
Brief Title: Effects of Atorvastatin 10 mg Versus 40 mg in Eight Months Follow-up Coronary Flow Reserve and Bone Marrow Stem Cell Mobilization in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Associate professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFR
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 10 mg versus 40 mg during the 8 months of follow-up

SUMMARY:
Many data indicate that statins increase mobilization of bone marrow-derived stem cells, and circulating bone marrow-derived stem cells are capable of homing to sites of myocardial infarction and endothelial disruption, thereby restoring myocardial function and microvascular integrity after acute myocardial infarction. Atorvastatin is widely used in the treatment of hyperlipidemia, especially after acute myocardial infarction. High-dose atorvastatin has been known to stop the progression of atherosclerosis and to decrease the levels of inflammatory markers.

The purpose of this prospective, randomized, single-blinded trial is to compare the effect of atorvastatin 10 mg versus 40 mg in restoring coronary flow reserve (CFR) and in serial bone marrow stem cell mobilization during the 8 months follow-up in patients with acute myocardial infarction.

DETAILED DESCRIPTION:
Percutaneous coronary intervention is considered as the gold standard for primary treatment after acute myocardial infarction, and clinical outcome and recovery of myocardial contractility after successful coronary intervention are influenced by the extent of microvascular damage. The use of intracoronary Doppler evaluation of infarct-related coronary artery allows direct assessment of microvascular integrity after acute myocardial infarction. The assessment of coronary flow reserve should be performed at least 24 hours after acute myocardial infarction, and we will evaluate coronary flow reserve 5 days after acute myocardial infarction. Intracoronary Doppler wire will be placed just distal to the stent, and intracoronary Doppler assessment is repeated 8 months after coronary stenting at the same point.

1. Primary end point: Comparison of atorvastatin 10 mg versus 40 mg on 8 months follow-up coronary flow reserve (CFR) and on the serial changes in stem cell mobilization (CD34, CD117, CD133, CXCR4+, C-met) after acute myocardial infarction.
2. Secondary end point: Comparison of atorvastatin 10 mg versus 40 mg on the changes in the levels of inflammatory markers (hsCRP, IL-6, TNF-α, adiponectin) and on the clinical events such as cardiac death, myocardial infarction, target vessel revascularization during the 8 months of follow-up.

1) Study design

* Prospective, randomized, single-blinded study.
* Patients enrollment: 100 patients (50 patients in each group) considering 20% drop-out rate.
* After informed consent, patients will be randomly assigned to the Atorvastatin 10 mg Group or the Atorvastatin 40 mg Group.

  2) Study protocol
* After IRB approval, we will enroll within 10 months 100 acute myocardial infarction patients requiring stent implantation.
* Study follow-up period will be 8 months.
* Baseline clinical, laboratory, and angiographic parameters will be obtained at baseline and at 8 months follow-up. Out-patients follow-up will be scheduled at 4 weeks, 16 weeks, 32 weeks after sirolimus-eluting stent implantation.
* We will compare atorvastatin 10 mg versus atorvastatin 40 mg on the changes in coronary flow reserve during the 8 months of follow-up. The serial changes (baseline, 24 hours, 48 hours, 5 days, 8 months) in stem cell mobilization (CD34, CD117, CD133, CXCR4+, C-met) will be compared in addition to major adverse cardiac events (cardiac death, myocardial infarction, target vessel revascularization) and inflammatory markers (hsCRP, IL-6, TNF-α, adiponectin).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Gender eligible for study both
* Patients with acute myocardial infarction requiring sirolimus-eluting stent implantation
* Acute myocardial infarction affecting proximal to mid coronary arteries
* No lesions greater than 50 percent diameter stenosis distal to the stent implantation
* Patients with informed consent

Exclusion Criteria:

* Left main lesion
* Killip Class IV acute myocardial infarction
* Patients with current use of any statin
* Tortuous lesion with difficult intracoronary Doppler wiring
* Acute myocardial infarction affecting distal coronary arteries
* Acute myocardial infarction affecting branching coronary arteries
* The use of thiazolidinediones within 3 months
* Previous history of PCI or bypass surgery on infarct-related coronary artery
* Patients with any contraindications to the treatment of atorvastatin
* Pregnant or lactating patients
* Chronic alcohol or drug abuse
* Hepatic dysfunction (3 times above upper normal limit 5 days after AMI)
* Renal dysfunction (Creatinine greater than 2.0 mg/dL)
* Severe Heart failure (EF less than 25 percent)
* Expected life expectancy of less thna 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Comparison of atorvastatin 10 mg versus 40 mg on 8 months follow-up coronary flow reserve (CFR) and on the serial changes in stem cell mobilization (CD34, CD117, CD133, CXCR4+, C-met) after acute myocardial infarction. | 8 month follow-up

SECONDARY OUTCOMES:
Comparison of atorvastatin 10 mg versus 40 mg on the changes in the levels of inflammatory markers (hsCRP, IL-6, TNF-α, adiponectin) and on the clinical events such as cardiac death, myocardial infarction, target vessel revascularization during the 8 mon | 8 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Soon Jun Hong, MD, PhD, Principal Investigator — Korea University Anam Hospital; Sang Yup Lim, MD, PhD, Study Director — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Hong SJ, Choi SC, Kim JS, Shim WJ, Park SM, Ahn CM, Park JH, Kim YH, Lim DS. Low-dose versus moderate-dose atorvastatin after acute myocardial infarction: 8-month effects on coronary flow reserve and angiogenic cell mobilisation. Heart. 2010 May;96(10):756-64. doi: 10.1136/hrt.2009.182683. PMID 20448126